CLINICAL TRIAL: NCT02165254
Title: Development of A Tai-Chi Program To Overcome Barriers To Cardiac Rehabilitation
Brief Title: The Gentle Cardiac Rehabilitation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Elena Salmoirago-Blotcher, Assistant Professor of Medicine, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34AT007569 (NIH); R34AT007569 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Secondary Prevention of Coronary Heart Disease
Keywords: physical activity; coronary heart disease; exercise; affect; mind/body therapies; stress, psychological
MeSH Terms: conditions — Motor Activity; Coronary Disease; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dose tai chi intervention (Other)
  Interventions: Behavioral: PLUS
- standard dose tai chi intervention (Other)
  Interventions: Behavioral: LITE

INTERVENTIONS:
Behavioral: PLUS — 1 hour tai chi session 3 times a week (weeks 1-12), to twice a week (week 13-16), and every other week (week 17-26) for a total of 24 weeks
  Arms: high dose tai chi intervention
Behavioral: LITE — 1 hour tai chi session 3 times a week (weeks 1-12)
  Arms: standard dose tai chi intervention

SUMMARY:
The purpose of this study is to develop a tai-chi based exercise program designed for patients who recently had a heart attack and do not wish, or are unable, to attend traditional cardiac rehabilitation.

DETAILED DESCRIPTION:
We will estimate the feasibility, acceptability and safety of two different doses of the Tai Chi intervention (primary outcome). 60 patients (30 per dose arm) will be randomly assigned to a standard dose of Tai Chi (the dose used by our group in large studies of heart failure patients) or to a high dose matching the recommended frequency and duration of exercise classes in current CRs. Acceptability assessments will include surveys and focus groups to formally assess the impact of Tai Chi on facilitators and barriers to CRs in this population. We will also obtain estimates of effect sizes of each dose on accelerometry measured physical activity and on the proportion of patients achieving the current American Heart Association (AHA) recommendation for physical activity (secondary outcome). Additional outcomes will be cardiac fitness, quality of life, body weight, and sleep. In addition, we will gather exploratory information on possible mechanisms by which Tai Chi training may affect physical activity. We will collect information on possible mediators such as exercise self-efficacy, perceived social support, and depression. In addition, since Tai Chi training is associated with meditative practices aimed at increasing present-moment awareness, we will gather information on mindfulness levels. Measurements will be conducted at baseline, 3-, 6-, and 9 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and speak English
2. Age ≥21
3. Physically inactive
4. Ability to understand the study procedures and willingness to commit to the demands of the study protocol

Exclusion Criteria:

1. Inability or unwillingness to give informed consent
2. Planning to move out of the area within the study period
3. Unstable angina
4. Blood pressure >200/110 or symptomatic orthostatic blood pressure decrease>20 mmHg
5. Uncontrolled atrial or ventricular arrhythmias; 3rd degree Atrio-Ventricular block
6. Pericarditis or myocarditis
7. Recent embolism/thrombophlebitis
8. Abnormal stress test without study cardiologist's clearance
9. Medical conditions likely to limit lifespan
10. NYHA functional class IV
11. Signs of cognitive impairment (BOMC >10)
12. Orthopedic problems prohibiting Tai Chi practice
13. Ongoing Tai Chi or other mind-body training
14. Current enrollment in a CR program
15. Severe depression (HADS scores>14)
16. Current drug or alcohol use or dependence that would interfere with adherence to study requirements.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
retention rates | up to 9 months since enrollment
drop-out rates | up to 9 months since enrollment
tai chi class attendance rates | up to 6 months since enrollment
number of participants with severe and non severe adverse events | up to 9 months since enrollment
percentage of participants reporting intervention acceptability scores in highest quartile | 3, 6, and 9 months since enrollment

SECONDARY OUTCOMES:
Mean between-group difference in within-participant change from baseline physical activity (accelerometry counts) over time (3, 6, and 9 months from enrollment) | baseline, 3, 6, 9 months
  To estimate mean between-doses differences in physical activity (and other continuous secondary outcomes listed below), we will estimate multivariate linear mixed models for within-participant change since baseline as a function of dose group (high or low), time point (3, 6, and 9 months from enrollment, treated as a categorical variable to allow for non-linear trajectories), and their interaction. A statistically significant interaction indicates that between-group differences vary across time points.

OTHER OUTCOMES:
Mean between-group difference in within-participant change from baseline Short Form-36 quality of life scores over time (3, 6, and 9 months from enrollment) | baseline, 3,6, and 9 months
Mean between-group difference in within-participant change from baseline HADS depression scores over time (3, 6, and 9 months from enrollment) | baseline, 3, 6, and 9 months
change from baseline aerobic capacity (METs) | baseline and intervention completion
Mean between-group difference in within-participant change from baseline Pittsburg Sleep Quality Index scores over time (3, 6, and 9 months from enrollment) | baseline, 3,6,9 months
Mean between-group difference in within-participant change from baseline Five Facets of Mindfulness (FFM) scores over time (3, 6, and 9 months from enrollment) | baseline, 3,6, and 9 months
Mean between-group difference in within-participant change from baseline Multidimensional Scale of Perceived Social Support scores over time (3, 6, and 9 months from enrollment) | baseline, 3, 6, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Salmoirago-Blotcher, PhD, MD, Principal Investigator — The Miriam Hospital & Warren Alpert Medical School at Brown University
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Salmoirago-Blotcher E, Wayne P, Bock BC, Dunsiger S, Wu WC, Stabile L, Yeh G. Design and methods of the Gentle Cardiac Rehabilitation Study--A behavioral study of tai chi exercise for patients not attending cardiac rehabilitation. Contemp Clin Trials. 2015 Jul;43:243-51. doi: 10.1016/j.cct.2015.06.020. Epub 2015 Jun 24. PMID 26115880
- [Result] Salmoirago-Blotcher E, Wayne PM, Dunsiger S, Krol J, Breault C, Bock BC, Wu WC, Yeh GY. Tai Chi Is a Promising Exercise Option for Patients With Coronary Heart Disease Declining Cardiac Rehabilitation. J Am Heart Assoc. 2017 Oct 11;6(10):e006603. doi: 10.1161/JAHA.117.006603. PMID 29021268